CLINICAL TRIAL: NCT05978765
Title: Effect of Dynamic Cupping Versus Myofascial Release on Pain, Range of Motion and Functional Performance in Athletes With Non-specific Low Back Pain
Brief Title: Effect of Dynamic Cupping & Myofascial Release on Pain, ROM and Performance in Athletes With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0414 UMER
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Low Back Pain; Myofascial Pain; Back Strain
Keywords: Athletic Performance; Low back pain; Myofascial release; Range of motion
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inclinometer (Experimental): Inclinometer : An inclinometer is a sensor used to measure the magnitude of the inclination angle or deformation of any structure
  Interventions: Device: Dry Cupping; Other: Myofascial Release
- Back Pain Functional Scale (Experimental): a subjective scale used to measure the patient's physical function after low back pain
  Interventions: Device: Dry Cupping; Other: Myofascial Release
- Functional Mobility Scale (Experimental): has been constructed to classify functional mobility
  Interventions: Device: Dry Cupping; Other: Myofascial Release
- Numeric Pain Rating Scale (Experimental): A pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable
  Interventions: Device: Dry Cupping; Other: Myofascial Release

INTERVENTIONS:
Device: Dry Cupping — treated by using dynamic cupping. Heating pad will be applied for 10 minutes as a base treatment then olive oil or petroleum jelly will be applied and a cup will be placed, a vacuum will be created by using vacuum pump then the cup will be moved to and fro or in figure of 8 for 5 minutes.
Other: Myofascial Release — e treated by soft tissue myofascial release. Heating pad will be applied for 10 minutes as a base treatment,petroleum jelly will be applied to the area follow by soft tissue myofascial release technique for 5 minutes either criss cross, along the fiber or in figure of 8

SUMMARY:
Data will be collected at Pakistan Sports Board Lahore. Study design will be Randomized Clinical Trial. Sample size is 28. Population will be divided into two Groups by Convinient Sampling Technique. Group A willl be Treated with Dynamic Cupping And Group B will be Treated with Soft Tissue Myofascial Release. Inclinometer, Back Pain Functional Scale, Functional Mobility Scale and Numerc Pain Rating Scale will be used to generate the outcomes of study.

DETAILED DESCRIPTION:
The objective of this study is to compare the Effects Of Dynamic Cupping Versus Myofascial Release on Pain, Range of motion and Function in athletes with non-specific low back pain.

Tools to be used in this study will be :

Inclinometer: An inclinometer is a sensor used to measure the magnitude of the inclination angle or deformation of any structure

. Back Pain Functional Scale: a subjective scale used to measure the patient's physical function after low back pain.

FMS: The Functional Mobility Scale (FMS) has been constructed to classify functional mobility.

Numeric PAIN Ratig Scale: The numeric rating scale (NRS) is a pain the screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".

The study will be collected from Sports related persons at Pakistan Sports Board Lahore. First, a consent form will be filled the person and then the data will be recorded through our questionaire on day 1 and then after 6 weeks of treatment. Group A will be treated with Dynamic Cupping and Group B will be treated with Myofascial release. Group A: will be an interventional group and it will be treated by using dynamic cupping. Heating pad will be applied for 10 minutes as a base treatment then olive oil or petroleum jelly will be applied and cup will be placed,a vacuum will be created by using a vacuum pump then the cup will be moved to and fro or in figure of 8 for 5 minutes. Group B : Will be a control group and it will be treated by soft tissue myofascial release. Heating pad will be applied for 10 minutes as a base treatment, and petroleum jelly will be applied to the area followed by soft tissue myofascial release technique for 5 minutes either crisscross, along the fiber or in Figure of 8.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* 18-35years(1)
* low Backpain
* NPRS (3 to 10 cut of value)
* Must be a Sports related persons.

Exclusion Criteria:

* Systemic Illness. (Diabetes mellitus,Tuberculosis, Arthritis, Scoliosis)
* History of Fracture in last 6 months
* Stayed out of Sports from last 6 months
* History of Disc Buldge and another structural problem.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Inclinometer | 10 months
  An inclinometer is a sensor used to measure the magnitude of the inclination angle or deformation of any structure
Back Pain Functional Scale | 10 Months
  a subjective scale used to measure the patient's physical function after low back pain
Functional Mobility Scale | 10 months
  The Functional Mobility Scale (FMS) has been constructed to classify functional mobility
Numeric Pain Rating Scale | 10 months
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable(

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohr C, Medina-Porqueres I. Immediate effects of myofascial release on neuromechanical characteristics in female and male patients with low back pain and healthy controls as assessed by tensiomyography. A controlled matched-pair study. Clin Biomech (Bristol). 2021 Apr;84:105351. doi: 10.1016/j.clinbiomech.2021.105351. Epub 2021 Apr 5. PMID 33848704
- [Background] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187
- [Background] Quinones S, Konschake M, Aguilar LL, Simon C, Aragones P, Hernandez LM, Abramovic A, Tubbs RS, Bouzada J, Valderrama-Canales FJ, Vazquez T, Sanudo J. Clinical anatomy of the lumbar sinuvertebral nerve with regard to discogenic low back pain and review of literature. Eur Spine J. 2021 Oct;30(10):2999-3008. doi: 10.1007/s00586-021-06886-1. Epub 2021 May 30. PMID 34052894
- [Background] Frost BA, Camarero-Espinosa S, Foster EJ. Materials for the Spine: Anatomy, Problems, and Solutions. Materials (Basel). 2019 Jan 14;12(2):253. doi: 10.3390/ma12020253. PMID 30646556
- [Background] Ughreja RA, Venkatesan P, Balebail Gopalakrishna D, Singh YP. Effectiveness of myofascial release on pain, sleep, and quality of life in patients with fibromyalgia syndrome: A systematic review. Complement Ther Clin Pract. 2021 Nov;45:101477. doi: 10.1016/j.ctcp.2021.101477. Epub 2021 Aug 27. PMID 34507243
- [Background] Salemi MM, Gomes VMDSA, Bezerra LMR, Melo TMS, Alencar GG, Montenegro IHPM, Calado APM, Montenegro EJN, Siqueira GR. Effect of Dry Cupping Therapy on Pain and Functional Disability in Persistent Non-Specific Low Back Pain: A Randomized Controlled Clinical Trial. J Acupunct Meridian Stud. 2021 Dec 31;14(6):219-230. doi: 10.51507/j.jams.2021.14.6.219. PMID 35770601
- [Background] Skelly AC, Chou R, Dettori JR, Turner JA, Friedly JL, Rundell SD, Fu R, Brodt ED, Wasson N, Kantner S, Ferguson AJR. Noninvasive Nonpharmacological Treatment for Chronic Pain: A Systematic Review Update [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2020 Apr. Report No.: 20-EHC009. Available from http://www.ncbi.nlm.nih.gov/books/NBK556229/ PMID 32338846
- [Background] Wang YT, Qi Y, Tang FY, Li FM, Li QH, Xu CP, Xie GP, Sun HT. The effect of cupping therapy for low back pain: A meta-analysis based on existing randomized controlled trials. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1187-1195. doi: 10.3233/BMR-169736. PMID 28946531
- [Background] Moura CC, Chaves ECL, Cardoso ACLR, Nogueira DA, Correa HP, Chianca TCM. Cupping therapy and chronic back pain: systematic review and meta-analysis. Rev Lat Am Enfermagem. 2018 Nov 14;26:e3094. doi: 10.1590/1518-8345.2888.3094. PMID 30462793
- [Background] Silva HJA, Saragiotto BT, Silva RS, Lins CAA, de Souza MC. Dry cupping in the treatment of individuals with non-specific chronic low back pain: a protocol for a placebo-controlled, randomised, double-blind study. BMJ Open. 2019 Dec 22;9(12):e032416. doi: 10.1136/bmjopen-2019-032416. PMID 31871257
- [Background] Rahyussalim AJ, Zufar MLL, Kurniawati T. Significance of the Association between Disc Degeneration Changes on Imaging and Low Back Pain: A Review Article. Asian Spine J. 2020 Apr;14(2):245-257. doi: 10.31616/asj.2019.0046. Epub 2019 Nov 5. PMID 31679325
- [Background] Oiestad BE, Hilde G, Tveter AT, Peat GG, Thomas MJ, Dunn KM, Grotle M. Risk factors for episodes of back pain in emerging adults. A systematic review. Eur J Pain. 2020 Jan;24(1):19-38. doi: 10.1002/ejp.1474. Epub 2019 Sep 3. PMID 31433541
- [Background] Sassack B, Carrier JD. Anatomy, Back, Lumbar Spine. 2023 Aug 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557616/ PMID 32491548
- [Background] Will JS, Bury DC, Miller JA. Mechanical Low Back Pain. Am Fam Physician. 2018 Oct 1;98(7):421-428. PMID 30252425
- [Background] Brandl A, Egner C, Schleip R. Reply to Kudus, A.L. Comment on "Brandl et al. Immediate Effects of Myofascial Release on the Thoracolumbar Fascia and Osteopathic Treatment for Acute Low Back Pain on Spine Shape Parameters: A Randomized, Placebo-Controlled Trial. Life 2021, 11, 845". Life (Basel). 2022 Jun 10;12(6):868. doi: 10.3390/life12060868. PMID 35743899
- [Background] Warren AJ, LaCross Z, Volberding JL, O'Brien MS. ACUTE OUTCOMES OF MYOFASCIAL DECOMPRESSION (CUPPING THERAPY) COMPARED TO SELF-MYOFASCIAL RELEASE ON HAMSTRING PATHOLOGY AFTER A SINGLE TREATMENT. Int J Sports Phys Ther. 2020 Aug;15(4):579-592. PMID 33354391
- [Background] Wood S, Fryer G, Tan LLF, Cleary C. Dry cupping for musculoskeletal pain and range of motion: A systematic review and meta-analysis. J Bodyw Mov Ther. 2020 Oct;24(4):503-518. doi: 10.1016/j.jbmt.2020.06.024. Epub 2020 Jul 30. PMID 33218554
- [Background] Kameda M, Tanimae H. Effectiveness of active soft tissue release and trigger point block for the diagnosis and treatment of low back and leg pain of predominantly gluteus medius origin: a report of 115 cases. J Phys Ther Sci. 2019 Feb;31(2):141-148. doi: 10.1589/jpts.31.141. Epub 2019 Feb 7. PMID 30858653
- [Background] Wu Z, Wang Y, Ye X, Chen Z, Zhou R, Ye Z, Huang J, Zhu Y, Chen G, Xu X. Myofascial Release for Chronic Low Back Pain: A Systematic Review and Meta-Analysis. Front Med (Lausanne). 2021 Jul 28;8:697986. doi: 10.3389/fmed.2021.697986. eCollection 2021. PMID 34395477
- [Background] Chen Z, Wu J, Wang X, Wu J, Ren Z. The effects of myofascial release technique for patients with low back pain: A systematic review and meta-analysis. Complement Ther Med. 2021 Jun;59:102737. doi: 10.1016/j.ctim.2021.102737. Epub 2021 May 10. PMID 33984499
- [Background] Liu YW, Su YL, Chang CL, Tsai MY. Cupping Therapy as an Adjunctive Therapy for Side Effects of Colorectal Cancer Treatment: A Prospective Observational Study. J Chiropr Med. 2022 Dec;21(4):280-287. doi: 10.1016/j.jcm.2022.02.011. Epub 2022 May 21. PMID 36420364